CLINICAL TRIAL: NCT00357812
Title: A Study to Compare the Efficacy of Two Potential Diagnostic Assays: a Fluorescein Conjugated Monoclonal Antibody in Vivo Assay and Nested Real Time PCR Assay to Rapidly and Accurately Diagnose Herpes Simplex Keratitis.
Brief Title: The Efficacy of Two Potential Diagnostic Assays for Herpes Simplex Keratitis (HSK)
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Bedford Hospital NHS Trust (Other); Midlands Eye Clinic (Unknown); Royal Victoria Hospital, Belfast (Other)
Other Study IDs: 04/NIR03/20
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-11

CONDITIONS: Herpes Simplex Keratitis
Keywords: Herpes Simplex Virus Type 1; Herpes Simplex Keratitis; Cornea; Dendretic Ulcer; In vivo Confocal Microscopy; Nested Multi-plex PCR; Monoclonal Antibody; Glycoprotein D; Glycoprotein C
MeSH Terms: conditions — Keratitis, Herpetic; Corneal Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The aim of this study is to compare the safety, specificity, sensitivity and ease of procedure of two potential diagnostic assays for HSV-1 detection in the cornea. Through the use of this new diagnostic assay, correct and early intervention would not only reduce corneal scarring from HSK, but it would also allow the initiation of appropriate treatment for HSV mimicking keratitis.

HSV-1 infection of the eye can result in corneal scarring and blindness. Early diagnosis of this condition and appropriate treatment is of utmost importance. Various ocular surface conditions can mimic herpetic keratitis in their clinical presentation and can result in diagnostic confusion. Inappropriate or delayed treatment of herpetic corneal disease results in increased morbidity.

In the UK at present clinical presentation is the mainstay of diagnosis. Unfortunately these cases often present to the most inexperienced clinical staff resulting in variability in diagnostic acumen. This often results in a delay or inappropriate diagnosis of herpetic keratitis. Laboratory techniques presently available to aid diagnosis are infrequently used in clinical practice. There are various reasons for their lack of use. Historically viral culture techniques were the mainstay of investigation but were slow, requiring weeks to provide a result. PCR is now replacing culture techniques and is relatively quick, reliable and sensitive. Many clinicians within the UK are still not fully informed of these advances and are therefore not utilizing these techniques to supplement clinical diagnosis.

We propose to investigate the use of topically applied fluorescent antibody against active replicating HSV-1 in a droplet form and real time PCR detection of the virus. If successful this should increase the potential diagnostic capabilities of GPs and other less experienced health care workers. Such tests should reduce variability in diagnosis and the dependency on experienced ophthalmologists to diagnose the condition.

DETAILED DESCRIPTION:
Strategy

Patients attending the Ophthalmology departments, who fulfil the criteria as outlined below in patient recruitment criteria, will be asked for written consent to volunteer for this study. Tears will be removed and stored in a sterile labelled eppendorf at -70 degrees C until further analysis. An impression cytology sample will be taken from the inflamed cornea and stored in viral transport medium and sent to the regional virology laboratory, Belfast for extraction and storage procedures. Blood samples will be taken and stored appropriately until the paired 3 month samples are available for antibody testing. Monoclonal antibody will be applied for the in vivo diagnosis of HSK as outlined below and viewed using an in vivo confocal microscope. Photographic evidence of the result will be recorded for each patient. Data for the nested real time PCR analysis and the monoclonal antibody test will be recorded separately by different individuals for each patient as the study progresses. Patient records will also be updated with the results of the tear and blood tests as the study progresses.

Recruitment Potential:

Over 200 eye patients in the RVH Belfast, over 300 patients in Bedford and over 600 patients in BMEC in Birmingham are treated each year with topical acyclovir for suspected HSV-1 infection. The number of patients treated within the community by GPs would significantly increase this number. The vast majority of these patients will have never had any laboratory confirmation of herpetic infection. The patient throughput through each hospital each year should enable adequate recruitment to this study over the three year period. This should ensure that the study is entirely viable from the perspective of patient numbers.

Patient numbers needed for a viable study

At present we are unable to perform statistical power calculations, as we are not aware of the sensitivity of either of the two proposed diagnostic assays. Previous work by Kaye SB20., et al has suggested a PCR technique with a sensitivity of 82% when used in human corneas). In contrast, the PCR technique used here should have a much superior sensitivity due to the use of real time analysis and the nested methodology used. These tests will be compared against the clinical diagnosis of an experienced consultant ophthalmologist.

We accept the need for statistical power calculations in order to calculate a recruitment level needed for a valid study. We will therefore carry out an initial study using all of these diagnostic assays on 50 patients and the results from this will be used to perform power calculations using the sample size method for one-sided equivalence of sensitivities based upon McNemar s test21 to ensure adequate numbers are recruited. In addition, we hope to over recruit (20% above this required number) to allow for patient dropout from the study.

Patient Recruitment Criteria

Patients over the age of 16 years in which the cause of keratitis is difficult to diagnose and in which HSK has to be excluded will be enrolled for this study. Immunosuppressed patients including patients treated with systemic steroids will be excluded. All patients will be asked for verbal and written consent. All patients will continue to be followed according to clinical requirements. In addition to routine assessment additional clinical categorisation by the attending consultants into those patients thought to (a) have, and (b) not have, clinical evidence in keeping with herpetic infection will be recorded.

In vivo immunofluorescence diagnostic procedure

30 microlitres of fluorescent-labelled mAB (2mg/ml), (same mAB as used in the previous study by Sharma A., et al7) in normal saline solution will be applied to the eye. After 20 minutes unbound antibody will be rinsed away with saline solution. The eye will be viewed with a slit lamp or an in vivo confocal microscope if available. mAB penetration through the layers of the cornea will be recorded. In addition, evidence of stromal inflammation will be recorded and its relationship to specific fluorescence noted. This will indicate the contribution of active herpetic infection (by specific fluorescence in either epithelium, stroma or both) as a causative effect rather than an immunological response to latent virus.

Comparison of in vivo results with nested real time PCR technique

Impression cytology will be carried out, prior to the application of the antibody, to confirm the presence/absence of viral antigens using nested real time PCR analysis. The potential for amplicon contamination associated with nucleic acid amplification test use is well recognised and makes mandatory the use of (a) separate, designated work stations and (b) a uni-directional work-flow from specimen preparation to amplified product analysis; this model of operation is standard in the regional virology laboratory. All PCR experiments will therefore be carried out under the supervision of Dr. Hugh O'Neill in the Regional Virology Laboratory, RVH, Belfast.

Impression cytology samples will be sent to the laboratory in viral transport medium. Each specimen will be vortexed for 15 seconds on receipt in the laboratory to resuspend the cellular content. A volume will be removed for PCR and the remainder will be stored.

Nested PCR will be undertaken using primers recognising the HSV-1 gpD gene (HSV-1 outer products will be 221 and 184 base pairs (bp) while the inner products will be 138 and 101 bp respectively). Hot-start PCR will be performed in a Perkin Elmer GeneAmp 2400 thermal cycler with 10 μl specimen plus 40 μl of mix and subjected to 35 first round cycles. One microlitre of product will be transferred to 49μl of second round mix for 25 second round cycles. Impression cytology samples taken from non-inflamed eyes from recruits with no history of herpetic eye infection will be used as known negative samples. A positive HSV control and a distilled water negative control will also be included in each run. First and second round products will be visualised together on ethidium bromide-stained 2% agarose gels and photographed (Polaroid). Appropriately sized bands present on second round only, or present on both first and second rounds, will be recorded as positive and strong positive respectively. All positive specimens will be re-tested.

Laboratory staff responsible for the PCR test will not be aware of the results from the in vivo antibody test. Comparison will be made between the sensitivity and specificity of the monoclonal antibody in vivo assay and the nested real time PCR diagnosis.

Investigating the effect of mAB on the ocular surface inflammatory milieu Analysis of the general cytokine profile will also be assessed by monitoring the cytokine profile of tears at two different time points: prior to monoclonal antibody treatment and again 30 minutes after the application of the antibody. Cytokine profile of tears will be analysed using proteomics with a protein biochip (RANDOX Labs. Ltd.) capable of simultaneous quantitative detection of an array of pro- and anti- inflammatory cytokines. Tear samples from patients suspected of active herpetic infection but who have not received antibody will serve as controls. Such analysis will allow statements to be made regarding the potential inflammatory/immunological reaction to the monoclonal antibody.

Investigating a potential systemic immunological reaction the mouse mAB Ten millilitres of clotted blood will be taken prior to the application of the monoclonal antibody to test for the presence of pre-existing antibody. In addition, at the 3 month check up a further 10 millilitres of blood will be taken and analysed again for antibodies which may have formed in the three month interface after the application of the monoclonal to the cornea.

The avascular cornea is thought to be an immunologically privileged site, making the potential of an immune response to the antibody less likely.

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 16 years in which the cause of keratitis is difficult to diagnose and in which HSK has to be excluded will be enrolled for this study

Exclusion Criteria:

Immunosuppressed patients including patients treated with systemic steroids will be excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients over the age of 16 years in which the cause of keratitis is difficult to diagnose and in which HSK has to be excluded will be enrolled for this study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Moore, PhD, Principal Investigator — Department of Biomedical Sciences, University of Ulster
Locations (3):
- United Kingdom (3):
  - Birmingham and Midlands Eye Clinic, Birmingham, Midlands
  - Bedford Hospital Ophthalmology Department and Acute Eye Clinic, Bedford
  - Royal Victoria Hospital, Belfast